CLINICAL TRIAL: NCT05311293
Title: Study on the Molecular Mechanism of Diarrhea-predominant Irritable Bowel Syndrome With Anxiety and Depression Based on Multi-omics Correlation Analysis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: irritable bowel syndrome
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with simple diarrhea-predominant irritable bowel syndrome
  Interventions: Diagnostic Test: Endoscopy
- Patients with irritable bowel syndrome accompanied by anxiety and depression
  Interventions: Diagnostic Test: Endoscopy
- Healthy Volunteers
  Interventions: Diagnostic Test: Endoscopy

INTERVENTIONS:
Diagnostic Test: Endoscopy — Observe the extent of colonic lesions and obtain intestinal mucosal samples

SUMMARY:
The research group intends to carry out a case-control study to recruit IBS-D patients with anxiety and depression symptoms, by collecting intestinal mucosa for single-cell transcriptome sequencing, collecting peripheral blood for proteomic analysis, the two groups and patient symptoms are associated, and then discover the characteristics of molecular level changes associated with brain-gut axis dysfunction, explore the pathophysiological mechanism of comorbid anxiety and depression and IBS, and discover potential targets for effective treatment. This project can help to construct the colonic single-cell map of IBS-D patients and explore the differentially expressed genes in the colon of IBS patients and their signaling pathways related to neuroregulation, providing an effective therapeutic target for the treatment of comorbid anxiety and depression and IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Rome IV diagnostic criteria for diarrhea-predominant irritable bowel syndrome;
2. Aged between 18 and 65 years old (inclusive), male or female;
3. HAMA assessment ≥ 14 points or HAMD assessment ≥ 17 points

Exclusion Criteria:

1. Patients with severe cardiovascular and cerebrovascular diseases (such as myocardial infarction, cerebral infarction, coronary heart disease, etc.);
2. Abnormal liver and kidney function (ALT or AST > 1.5 times the upper limit of normal, or T-Bil > 1.5 times the upper limit of normal, or Cr more than the upper limit of normal), hematopoietic system diseases and tumors;
3. Patients with a history of abdominal surgery (except appendectomy and cholecystectomy);
4. Previous diagnosis of organic diseases of the digestive system, such as inflammatory bowel disease, intestinal tuberculosis, etc., or still associated with peptic ulcer, infectious diarrhea, etc.;
5. Previous diagnosis of diseases similar to irritable bowel syndrome symptoms, such as eosinophilic enteritis, microscopic colitis (including collagen colitis and lymphocytic colitis), lactose intolerance, malabsorption syndrome;
6. Previous diagnosis of non-intestinal digestive system diseases, such as tuberculous peritonitis, gallstones, cirrhosis, chronic pancreatitis;
7. Previous diagnosis of diseases affecting the digestive tract function, such as hyperthyroidism or hypothyroidism, endometriosis, autoimmune diseases, diabetes, etc.;
8. 4. Patients who have taken drugs with bleeding risk or increased bleeding risk before treatment;
9. 4. Patients who have taken antidepressant drugs and psychotropic drugs before treatment;
10. 4. Use drugs that affect gastrointestinal motility and function, such as prokinetic drugs, anticholinergic drugs, calcium channel blockers, 5-HT receptor agonists/antagonists, antidiarrheal agents, antacids, intestinal bacteria modulators and antibiotics;
11. Allergic constitution;
12. Pregnant and lactating women; Others that may affect study compliance or adversely affect the results as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Meet the Rome IV diagnostic criteria for diarrhea-predominant irritable bowel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Depression Score | up to 100 weeks
  To evaluate the extent to which a disease affects a mental condition

CONTACTS AND LOCATIONS:
Locations (1):
- Tang-Du Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: Undecided